CLINICAL TRIAL: NCT03617484
Title: Phase II Study Evaluating the Effect of Adding Bortezomib to Ibrutinib in Ibrutinib Relapsed Mantle Cell Lymphoma
Brief Title: Bortezomib in Combination With Ibrutinib in Ibrutinib Relapsed Mantle Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment and/or interactions/interventions temporarily paused due to COVID-19 and expected to resume in the future. This is not a suspension of IRB approval.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.046; HUM00139543 (Other: University of Michigan)
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Mantle Cell Lymphoma
Keywords: Relapsed
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — Bortezomib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bortezomib + Ibrutinib (Experimental): Ibrutinib will be administered orally at a dose of 560 mg daily for each 21 day cycle.
  Bortezomib will be administered subcutaneously at a dose of 1.3 mg/m^2 on days 1, 4, 8, and 11 of each 21-day cycle.
  Interventions: Drug: Bortezomib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be administered subcutaneously at a dose of 1.3 mg/m^2 on days 1, 4, 8, and 11 of each 21-day cycle.
Drug: Ibrutinib — Ibrutinib will be administered orally at a dose of 560 mg daily for each 21 day cycle.

SUMMARY:
This is a phase II study to evaluate the efficacy of ibrutinib in combination with bortezomib in in MCL (mantle cell lymphoma) patients who relapsed on single agent ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Diagnosis of mantle cell lymphoma established by histologic assessment by a hemato-pathologist with additional assessment of the histologic diagnosis by immunohistochemistry or flow cytometry.
* Patients with history of MCL that has relapsed (documented disease progression after previously responding) to therapy (CR/PR) on single agent ibrutinib (treated for at least 6 months) as the last treatment prior to enrollment.
* Adequate liver, renal and bone marrow function
* Adequate coagulation (unless abnormalities are unrelated to coagulopathy or bleeding disorder)
* Female subjects of childbearing potential must have a negative urine/serum pregnancy test upon study entry. Women as well are not advised to breastfeed during treatment with bortezomib and for 2 months after treatment.
* Male and female subjects of reproductive potential must agree to use both a highly effective method of birth control and barrier method during the period of therapy and for 30 days after the last dose of study drug for females and 90 days for males.
* Eastern Cooperative Oncology Group (ECOG) performance status of <2 (Eastern Cooperative Oncology Group scoring system used to quantify general well-being and activities of daily life; scores range from 0 to 5 where 0 represents perfect health and 5 represents death.)

Exclusion Criteria:

* Concurrent diagnosis of another malignancy unless treated with curative intent more than 2 years from study start (basal/squamous cell carcinoma of the skin is not an exclusion).
* Previous treatment with bortezomib.
* Patients who are eligible for autologous stem cell transplant are excluded unless they refuse this procedure.
* History of allogeneic stem cell transplant.
* Other exclusions (certain concurrent conditions) per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants that respond to treatment at 6 months | 6 Months
  The primary endpoint is overall response rate (ORR). Participants will be evaluated for response based on the Lugano criteria.

SECONDARY OUTCOMES:
Overall survival time | Up to 10 Years
  Patients will be followed for survival until death or up to 10 years.
Progression free survival time | Up to 10 Years
  Progression will be determined using the Lugano criteria. Patients will be followed for survival until death or up to 10 years.
Best overall response | Up to 10 Years
  Participants will be evaluated for response based on the Lugano criteria. From the start of the study treatment until the disease progression/recurrence or up to 10 years.
Rate of complete response | Up to 10 Years
  Participants will be evaluated for response based on the Lugano criteria. The percentage of participants who achieve CR after treatment.
Time to progression | Up to 10 Years
  Progression will be determined using the Lugano criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tycel Phillips, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No